CLINICAL TRIAL: NCT04658979
Title: Evaluation of the Feasibility and Safety of a Pulmonary Tele-rehabilitation Program in the Times of COVID-19
Brief Title: Pulmonary TELE-REHABilitation Program : Feasibility and Safety Study
Acronym: Tele-RehaB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Collaborators: Fondation IUCPQ (Other)
Responsible Party: Principal Investigator, Didier Saey, Principal investigator, Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21983
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Chronic Pulmonary Disease
Keywords: Pulmonary Telerehabilitation; Safety; Feasibility; Interstitial lung disease; Chronic obstructive lung disease
MeSH Terms: conditions — Lung Diseases, Interstitial; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental)
  Interventions: Other: Pulmonary tele-rehabilitation

INTERVENTIONS:
Other: Pulmonary tele-rehabilitation — All the participant will by include in a tele-rehabilitation program who will be based on an 12-week intervention including therapeutic education and self-management sessions and training sessions, delivered through a videoconferencing application. All interventions will be under the supervision of a rehabilitation professional from the Pavillon de prévention des maladies cardiovasculaire (PPMC) and modeled according to the recommendations of the ATS/ERS.

SUMMARY:
Chronic pulmonary disease like interstitial lung disease (ILD) and chronic obstructive lung disease (COPD) are a significant health problem in Canada and around the world. In addition to the respiratory impairment resulting to a progressive dyspnea, these diseases are also characterized by a decrease in exercise tolerance and muscle dysfunction which affect the patient's quality of life. Respiratory rehabilitation is the cornerstone of the management of chronic disease and it includes a set of personalized care mainly delivered in person by a transdisciplinary team and with the objectives of reducing the symptoms felt by the participants and improving their physical and psychosocial condition.

The current containment due to the COVID-19 pandemic increase the sedentary behavior of patients and prevents the holding of any respiratory rehabilitation activity. In this context, tele-rehabilitation appears to be a particularly well-suited solution because it would make it possible to offer a respiratory rehabilitation in a safe and effective manner while minimizing contact with the participants. Although some studies support the feasibility of this intervention, more data is needed to validate its routine clinical application.

The main objective of this study is to verify the safety and the feasibility of delivering pulmonary rehabilitation treatments entirely at home via a telerehabilitation patform developed at the Institut universitraire de cardiologie et de pneumologie de Québec (IUCPQ), and document its effectiveness in people with chronic respiratory disease. The secondary objectives will be: 1) to explore the effects of a telerehabilitation programm on exercise tolerance, muscle function, functional capacity and quality of life, and 2) to assess the satisfaction of participants and health care providers with telerehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* The patient already participate to the telerehabilitation program in the PPMC at IUCPQ

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Feasability - Patients´ satisfaction with the program between baseline and the up to 12 weeks follow-up | 12 weeks
  Patient's satisfaction will be evaluated by a questionnaire including 7 questions on his feeling of competence with regard to the program, based on an 8-point Likert scale (0 to 7).
Feasability - Health care professionals' receptivity | 12 weeks
  Health care professionals' receptivity towards the tele-rehabilitation will be assess by 18 questions based on an 6-point scale (0 to 5).
Feasibility - Patients' satisfaction with the health care received | 12 weeks
  Patient's satisfaction will be evaluated by a questionnaire including 23 questions based on a 4-point scale (1 to 4).

SECONDARY OUTCOMES:
Quality of life by questionnaire | 12 weeks
  For the COPD participants the quality of live will be evaluated with the COPD Assessment test (CAT) and fort he ILD participants with the Kings' Brief Interstitial Lung Disease (K-BLID) questionnaire.
  CAT = K-BLID = 15 questions rate between 1 to 7 (maximal score = 105 = better quality of life; minimal score = 15 = worse quality of life)
Dyspnea level | 12 weeks
  The dyspnea level will be evaluated with the MRC questionnaire = 4 questions If the patient answer yes to the first question he continue to the next question, if he answer no the questionnaire is finish. The further he goes in the questionnaire, worse the breathlessness score is.
Exercise capacity | 12 weeks
  The exercise capacity will be evaluated by the 6-minutes stepper test before and after the program, the result will be the number of cycle complet
Exercise capacity | 12 weeks
  The exercise capacity will be evaluated by the 1-minute sit to stand test before and after the program, the result will be the number of complet sit to stand.
Functionnal capacity | 12 weeks
  The functional capacity will be evaluated by the Short Physical Performance Battery test (SPPB) test before and after the program, the result will be the total on 12.
Functionnal capacity | 12 weeks
  The functional capacity will be evaluated by the hand grip test before and after the program and measured in kilograms.
Functionnal capacity | 12 weeks
  The functional capacity will be evaluated by the maximum voluntary contraction force of the quadriceps before and after the program.
Anxiety | 12 weeks
  The anxiety will be assess by the Hospital Anxiety and Depression scale (HAD). Total of 14 questions (maximal score = 42 = worse; minimal score = 0= better) where 7 questions is for the anxiety score(maximal score = 21 = worse; minimal score = 0= better)
Depression | 12 weeks
  The depression will by assess by Hospital Anxiety and Depression scale.14 questions (maximal score = 42 = worse; minimal score = 0= better) where 7 questions is for the depression score (maximal score = 21 = worse; minimal score = 0= better)

CONTACTS AND LOCATIONS:
Overall Officials: Didier Saey, Ph.D, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec -ULaval
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada